CLINICAL TRIAL: NCT01308021
Title: Clinical Efficacy, Immunogenicity, Clinical Tolerability and Assessment of Safety of gpASIT+TM Administered Orally, According to Two Administration Schedules, for the Prophylaxis of Seasonal Grass Pollen Rhinoconjunctivitis
Brief Title: Clinical Efficacy and Safety of gpASIT+TM to Treat Seasonal Allergic Rhinoconjunctivitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BioTech Tools S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: BTT-gpASIT005
Record Dates: First submitted 2011-02-28; First posted 2011-03-03 (Estimated); Last update posted 2014-05-26 (Estimated); Status verified 2014-05

CONDITIONS: Grass Pollen Allergy; Hay Fever
Keywords: Rhinoconjunctivitis; Allergy; Grass pollen; Hypersensitivity; Immune system disorder
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal; Hypersensitivity; Immune System Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- gpASIT400 (Experimental): gpASIT+TM 400 µg
  Interventions: Biological: gpASIT+TM
- gpASIT800 (Experimental): gpASIT+TM 800 µg
  Interventions: Biological: gpASIT+TM
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: gpASIT+TM — entero-coated capsules containing 400µg of gpASIT+TM, daily , 28 days
  Arms: gpASIT400
Biological: gpASIT+TM — entero-coated capsules containing 800 µg of gpASIT+TM, daily, 28 days
  Arms: gpASIT800
Biological: Placebo — Placebo entero-coated capsules
  Arms: Placebo

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of grass pollen-derived peptides administrated orally to treat seasonal allergic rhinoconjunctivitis.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 50 years
* Subject has given written informed consent
* The subjects are in good physical and mental health according to his/her medical history, vital signs, and clinical status
* Male or non pregnant, non-lactating female
* Female unable to bear children must have documentation of such in the CRF (i.e. tubule ligation, hysterectomy, or post menopausal (defined as a minimum of one year since the last menstrual period))
* Allergy > 2 years

Exclusion Criteria:

* Subjects with current immunotherapy or subjects who underwent a previous immunotherapy within the last 2 years
* Subjects with perennial asthma
* Subjects with a VC < 80% and FEV1 < 70%
* Subjects requiring controller medication against asthma (bronchodilator nebulised drugs or local or systemic corticosteroids)
* Documented evidence of chronic sinusitis (as determined by investigator)
* Subjects with a history of hepatic or renal disease
* Subjects symptomatic to perennial inhalant allergens
* Subject with malignant disease, autoimmune disease
* Female subjects who are pregnant, lactating, or of child-bearing potential and not protected from pregnancy by a sufficiently reliable method (OCs, IUD, ...)
* Any chronic disease, which may impair the subject's ability to participate in the trial (i.e. severe congestive heart failure, active gastric ulcer, inflammatory bowel disease, uncontrolled diabetes mellitus, etc…)
* Subjects requiring beta-blockers medication
* Chronic use of concomitant medications that would affect assessment of the effectiveness of the trial medication (e.g. tricyclic antidepressants)
* Subject with febrile illness (> 37.5°C, oral)
* A known positive serology for HIV-1/2, HBV or HCV
* The subject is immunocompromised by medication or illness, has received a vaccine, corticoids or immunosuppressive medications within 1 month before trial entry
* Receipt of blood or a blood derivative in the past 6 months preceding trial entry
* Regular consumption of corticoids (oral, topic or nasal) or of anti-histaminic drugs within 4 weeks preceding the trial
* Any consumption of corticoids (oral, topic or nasal) or of anti-histaminic drugs within 1 week preceding the trial
* Use of long-acting antihistamines
* Any condition which could be incompatible with protocol understanding and compliance
* Subjects who have forfeited their freedom by administrative or legal award or who are under guardianship
* Unreliable subjects including non-compliant subjects, subjects with known alcoholism or drug abuse or with a history of a serious psychiatric disorder as well as subjects unwilling to give informed consent or to abide by the requirements of the protocol
* Participation in another clinical trial and/or treatment with an experimental drug within the last 2 years
* A history of hypersensitivity to the excipients
* Rhinitis medicamentosa, non-specific rhinitis (to food dye, preservative agent…)
* Subjects without means of contacting the investigator rapidly in case of emergency, or not able to be contacted rapidly by the investigator

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 202 (Actual)
Dates: Start 2010-12; Primary Completion 2011-10 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Impact of gpASIT+TM on the clinical efficacy of the subjects | grass pollen season 2011 (April to July)
  The following parameter will be assessed: rhinoconjunctivitis total symptom score

SECONDARY OUTCOMES:
Clinical tolerability and safety of the treatment | 8 months
  The following parameters will be assessed: general physical status, vital signs, haematological parameters, general blodd biochemistry parameters, all (serious) adverse events, immunological analysis (total IgG, IgE) and inflammatory parameters (CRP, sedimentation rate)
Impact of gpASIT+TM on the immunological status of the subjects | screening visit (January-February 2011), before pollen season (April 2011), during pollen season (June 2011) and after pollen season (August 2011)
  The following parameter will be assessed: allergen-specific immunoglobulin concentrations
Impact of gpASIT+TM on the clinical status of the subjects | grass pollen season 2011 (April-July)
  The average daily symptom and rescue medication scores will be assessed.
Impact of gpASIT+TM on the quality of life of the subjects | grass pollen season 2011 (April-July)
  The quality of life will be assessed by the use of validated questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Claus Bachert, MD, Principal Investigator — UZ Ghent; Jan Ceuppens, MD, Principal Investigator — UZ Leuven; Didier Ebo, MD, Principal Investigator — UZ Antwerpen; Jean-Luc Halloy, MD, Principal Investigator — CHR Warquignies; Stijn Hallewyck, MD, Principal Investigator — Universitair Ziekenhuis Brussel; Peter Hellings, MD, Principal Investigator — UZ Leuven; Renaud Louis, MD, Principal Investigator — Centre Hospitalier Universitaire de Liege; Catherine Mbasoa, MD, Principal Investigator — Clinique du Parc Léopold Bruxelles; Charles Pilette, MD, Principal Investigator — UCL Saint Luc Bruxelles; Hélène Simonis, MD, Principal Investigator — CHR Citadelle Liège; Olivier Vandenplas, MD, Principal Investigator — UCL Mont Godinne Yvoir; Christoph Verhoye, MD, Principal Investigator — AZ Sint-Lucas Brugge; Patricia Wackenier, MD, Principal Investigator — CHU Ambroise-Paré - Mons; Frédéric De Blay, MD, Principal Investigator — CHRU Strasbourg; Marie-Christine Castelain, MD, Principal Investigator — Hôpital Saint Vincent de Paul, Lille; François Lavaud, MD, Principal Investigator — CHRU Reims; Benoît Wallaert, MD, Principal Investigator — CHU Lille; François Wessel, MD, Principal Investigator — Private Practice Nantes; Bruno Lebeaupin, MD, Principal Investigator — Private Practice Nantes; François Hentges, MD, Principal Investigator — CHL Luxembourg; François Durand Perdriel, MD, Principal Investigator — Private Practice Nantes; François Spirlet, MD, Principal Investigator — CH de Dinant
Locations (18):
- Belgium (12):
  - CHR Saint Joseph Warquignies, Boussu
  - AZ Sint Lucas, Bruges
  - Clinique du Parc Léopold, Brussels
  - UZ Brussel, Brussels
  - UCL Saint Luc, Brussels
  - UZ Antwerpen, Edegem
  - UZ Gent, Ghent
  - UZ Leuven, Leuven
  - CHR Citadelle, Liège
  - CHU Sart-Tilman, Liège
  - CHU Ambroise Paré, Mons
  - UCL Mont Godinne, Yvoir
- France (5):
  - Hôpital Saint Vincent de Paul, Lille
  - CHRU Lille, Lille
  - Private practice, Nantes
  - CHU Reims, Reims
  - CHRU Strasbourg, Strasbourg
- CH Luxembourg, Luxembourg, Luxembourg